CLINICAL TRIAL: NCT05428397
Title: Safety Profile of Ultravist in Patients With Different Sexes, Races and From Different Countries/Regions
Brief Title: A Study, Called UV Population, to Learn More About the Safety of the Study Drug Ultravist, Which is Given to Get Clearer X-ray Pictures, in People of Different Sexes, Races, and From Different Countries/Regions
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22133
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Contrast Enhanced X-ray Based Examination
Keywords: Hypersensitivity reaction; CT; Angiography; Contrast enhancement; Computed tomography
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Contrast enhanced X-ray based examination with Ultravist: Patients who received a contrast enhanced X-ray based examination with Ultravist for various clinical reasons and having experienced a hypersensitivity reaction.
  Interventions: Diagnostic Test: Iopromide (Ultravist, BAY86-4877)
- Control group: Patient who received contrast enhanced X-ray based examination with Ultravist for various indications who had not adverse event.
  Interventions: Diagnostic Test: Iopromide (Ultravist, BAY86-4877)

INTERVENTIONS:
Diagnostic Test: Iopromide (Ultravist, BAY86-4877) — X-Ray/CT Diagnostic Imaging
  Other Names: BAY86-4877_Iopromide_IV_X-Ray/CT Diagnostic Agents

SUMMARY:
This is an observational study in which patient data from the past of people who received Ultravist prior to an X-ray based scan are studied.

In observational studies, only observations are made without specified advice or interventions.

X-ray based imaging like computed tomography or angiography is used to make pictures of the structures inside the body. These pictures are needed in various medical situations. In some X-ray tests, the patient is given a compound called "contrast agent" that is injected into the vein. It helps to create clearer pictures as it makes internal body structures easier to see. With such contrast-enhanced imaging techniques, doctors can better see certain problems.

Ultravist is an iodine-based contrast agent. It is also called iopromide, and it is available for doctors to give patients before they have X-ray based scans.

Clinical studies on the overall safety of Ultravist have shown that hypersensitivity reactions (HSRs) may rarely occur. HSRs are undesirable reactions of the body's defense system (immune system) to the study drug. However, more information on HSRs is needed.

The main aim of this study is to find out whether certain groups of people are more likely to have HSRs after Ultravist injection than others (e.g., depending on gender, race, or country/region).

To do this, researchers will collect data from people with HSRs (all ages) after contrast-enhanced X-ray scans with Ultravist. These data come from four observational studies that have already been completed. Participants who had HSRs will be compared with participants in these studies who had no medical problems after receiving Ultravist to learn more about the characteristics of people at higher risk.

Data will be from the year 1999 up to 2011. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all age groups which were referred to any iodine-based contrast-enhanced procedure after administration of either Ultravist 300 mg I/mL or 370 mg I/mL.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: In this integrated analysis, the data of four company sponsored non-interventional studies with Ultravist in contrast-enhanced X-ray examination have been pooled. This pool consists of studies 'PMS I', 'IMAGE', 'TRUST', 'Ultravist in CT'.The total data pool consists of 152,233 patients. The timeframe of these 4 studies is from 6/1999 until 11/2011. The study utilizes data collected as a part of clinical practice across 37 countries and including Europe (mostly Germany and Spain), Asia (mostly China and South Korea) and USA. It will not include any new and not yet published data. Patients of all ages, both sexes, multiple races and across various health conditions/indications are represented in this pooled database.
Sampling Method: Non-Probability Sample
Enrollment: 152233 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Hypersensitivity reaction (HSR) to Ultravist (iopromide) in patients with different sex | ≤1 hour after contrast administration
  Cases (based on MedDRA version 21.0): Patients with any typical and unequivocal hypersensitivity reaction: anaphylactoid shock, angioedema, asthma, bronchospasm, conjunctivitis, cough, dysphagia, dyspnea, edema mucosal, erythema/exanthema/rash, hoarseness, lacrimation, laryngeal/pharyngeal/face edema, laryngeal/pharyngeal spasm, nasal stuffiness, pruritus/itching, respiratory arrest, rhinitis, sneezing, stridor, swelling (eyes/face), throat irritation, tongue edema, urticaria/hives/blisters, wheezing.
Hypersensitivity reaction (HSR) to Ultravist (iopromide) in patients with different race | ≤1 hour after contrast administration
Hypersensitivity reaction (HSR) to Ultravist (iopromide) in patients from different countries/regions | ≤1 hour after contrast administration

SECONDARY OUTCOMES:
Differences regarding specific HSRs in patients with different sex | ≤1 hour after contrast administration
Differences regarding specific HSRs in patients with different race | ≤1 hour after contrast administration
Differences regarding specific HSRs in patients from different countries/regions | ≤1 hour after contrast administration

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer, Wuppertal, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Background] Palkowitsch P, Lengsfeld P, Stauch K, Heinsohn C, Kwon ST, Zhang SX, Liang CH. Safety and diagnostic image quality of iopromide: results of a large non-interventional observational study of European and Asian patients (IMAGE). Acta Radiol. 2012 Mar 1;53(2):179-86. doi: 10.1258/ar.2011.110359. Epub 2011 Dec 19. PMID 22184683
- [Background] Chen W, Mempel M, Schober W, Behrendt H, Ring J. Gender difference, sex hormones, and immediate type hypersensitivity reactions. Allergy. 2008 Nov;63(11):1418-27. doi: 10.1111/j.1398-9995.2008.01880.x. PMID 18925878
- [Background] Chen JY, Liu Y, Zhou YL, Tan N, Zhang B, Chen PY, Chen LB. Safety and tolerability of iopromide in patients undergoing cardiac catheterization: real-world multicenter experience with 17,513 patients from the TRUST trial. Int J Cardiovasc Imaging. 2015 Oct;31(7):1281-91. doi: 10.1007/s10554-015-0688-9. Epub 2015 Jun 10. PMID 26058857
- [Result] Kopp AF, Mortele KJ, Cho YD, Palkowitsch P, Bettmann MA, Claussen CD. Prevalence of acute reactions to iopromide: postmarketing surveillance study of 74,717 patients. Acta Radiol. 2008 Oct;49(8):902-11. doi: 10.1080/02841850802282811. PMID 18651252
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field — https://clinicaltrials.bayer.com